CLINICAL TRIAL: NCT03132961
Title: Effects of Infrasound Exposure on Measures of Endolymphatic Hydrops
Status: Terminated | Type: Observational
Why Stopped: Despite recruitment of healthy volunteers, participants from the population of interest were unable to be recruited.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1701M04145
Record Dates: First submitted 2017-03-09; First posted 2017-04-28 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Vestibular Abnormality; Endolymphatic Hydrops
Keywords: Vestibular evoked myogenic potentials; Electrocochleography; Infrasound
MeSH Terms: conditions — Endolymphatic Hydrops

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Block 1: Participants in the cohort will undergo testing in the order of: ECoG, oVEMP, cVEMP
  Interventions: Other: Infrasound exposure
- Block 2: Participants in the cohort will undergo testing in the order of: ECoG, cVEMP, oVEMP
  Interventions: Other: Infrasound exposure
- Block 3: Participants in the cohort will undergo testing in the order of: oVEMP, cVEMP, ECoG
  Interventions: Other: Infrasound exposure
- Block 4: Participants in the cohort will undergo testing in the order of: oVEMP, ECoG, cVEMP
  Interventions: Other: Infrasound exposure
- Block 5: Participants in the cohort will undergo testing in the order of: cVEMP, ECoG, oVEMP
  Interventions: Other: Infrasound exposure
- Block 6: Participants in the cohort will undergo testing in the order of: cVEMP, oVEMP, ECoG
  Interventions: Other: Infrasound exposure

INTERVENTIONS:
Other: Infrasound exposure — All cohorts will receive an identical infrasound exposure of equal time duration, varying only the order in which the testing is performed. To simulate the frequencies generated by a common source of environmental infrasound (wind turbines), recordings measured at a full-scale research wind turbine at the University of Minnesota will be utilized to create an infrasound stimulus. The resultant sound file consists of the fundamental frequency at approximately 0.7 Hz, equal to the blade passage rate, plus the harmonic overtones of the fundamental frequency. The presentation level is 85 dB SPL. The stimulus will be presented in a sound field.

SUMMARY:
Persons exposed to infrasound - frequencies below 20 Hz - describe a variety of troubling audiovestibular symptoms, but the underlying mechanisms are not understood. Recent animal studies, however, provide evidence that short-term exposure to low frequency sound induces transient endolymphatic hydrops. The existence of this effect has not been studied in humans. The long-term objective of this research is to identify a possible mechanism to describe the effects of infrasound on the human inner ear. The central hypothesis of the proposed study is that short-term infrasound exposure induces transient endolymphatic hydrops in humans. This will be tested by performing electrophysiologic tests indicative of endolymphatic hydrops among normal hearing individuals before and immediately after a period of infrasound exposure. Recordings of infrasound generated by wind turbines in the field have been established and calibrated by this team of engineers, otologist, and hearing and balance scientists. An infrasound generator reproduces the acoustic signature based on these field recordings. Aim 1: Determine the effect of infrasound on the summating potential to action potential (SP/AP) ratio on electrocochleography (ECoG). Hypothesis 1: Infrasound exposure will cause a reversible elevation of the SP/AP ratio. Aim 2: Determine the effect of infrasound on the threshold response curves of ocular and cervical vestibular evoked myogenic potentials. (oVEMP and cVEMP). Hypothesis 2: Infrasound exposure will cause elevation of the oVEMP and cVEMP thresholds at the frequency of best response. Successful completion of the aims will provide evidence for a possible mechanism of the effect of infrasound on the inner ear. This understanding will benefit individuals exposed to environmental infrasound and those in regulatory, research, and advocacy roles when crafting interventions and future policy.

DETAILED DESCRIPTION:
Infrasound is generated within the human body by processes such as respiration and myocardial contraction. External sources include those produced naturally, such as wind and earthquakes, and those that are human-made, such as automobile engines and heavy machinery. Wind turbines are known to emit infrasound with a fundamental frequency of 1 Hz with intensities approaching 100 decibels (dB), depending on wind speed. Over 75,000 wind turbines have been deployed between 2003 and 2015 in the U.S. alone. As environmental infrasound exposure has increased in prevalence and intensity with the advent of technologies such as large-scale wind turbines, renewed attention has been directed to the effects of infrasound on exposed individuals.

As it falls below audible thresholds, conventional wisdom would dictate that infrasound does not affect humans. However, some individuals living in proximity to wind turbines experience increased levels of annoyance and sleep disturbance in a dose-response fashion. Other reported symptoms from infrasound exposure include aural fullness, tinnitus, dizziness, and vertigo. Some researchers hypothesize that these otologic symptoms are related to the infrasonic component of wind turbine noise affecting inner ear function. However, since the mechanism or causal role have yet to be established, others attribute such symptoms to a psychosomatic or "nocebo" effect (i.e. worsening symptoms produced by negative expectations). As wind farms and other infrasound-generating sources become widespread, there is now a critical need to determine the effects of infrasound on inner ear function.

Studies conducted in humans have confirmed that infrasound has measurable effects within the cochlea. Hensel et al presented infrasound tones of 6 and 12 Hz at 130 dB sound pressure level (SPL) while simultaneously measuring distortion product otoacoustic emissions (DPOAEs). They observed considerable increases in DPOAE amplitudes in the presence of infrasound compared to when these tones were absent. The authors attributed this effect to the displacement of the cochlear partition during infrasound exposure. Further, Dommes et al demonstrated activity in the primary auditory cortex on functional magnetic resonance imaging during infrasound exposure, providing evidence that perception of infrasound occurs through known auditory pathways.

Reversible hydropic changes of the endolymphatic space have been observed during short-term exposure to infrasound and low frequency sound in several guinea pig models. Flock and Flock utilized an explanted guinea pig temporal bone model to visualize expansion of the endolymphatic space on confocal microscopy while applying tone bursts of 140 Hz between 88-112 dB. Shortly after this work, Salt detected changes indicative of endolymphatic hydrops in vivo using volume and flow markers iontophoresed into the endolymphatic space of guinea pigs during 3 minutes of exposure to 200 Hz tone bursts at 115 dB SPL. The observed changes in flow and volume in the endolymphatic space were reversible. The recovery half time in this study was 3.2 minutes. Subsequent work by Salt et al demonstrated that infrasound at 5 Hz generated larger endolymphatic potentials in the third cochlear turn than did frequencies in the audible range from 50-500 Hz. This was despite a presentation level expected to be below the hearing threshold of the guinea pigs. These studies demonstrate that infrasound and low-frequency tones have measurable effects on inner ear physiology, even at sub-threshold hearing levels.

While there is evidence that the human cochlea is stimulated by infrasound, it is not known if infrasound induces endolymphatic hydrops in humans. The proposed work will test the central hypothesis that short-term infrasound exposure induces reversible endolymphatic hydrops in the human inner ear. This hypothesis is based on the observations in the presented animal studies and the observed combination of auditory and vestibular symptoms reported to be associated with infrasound exposure.

In order to test the hypothesis in living humans, the proposed study will utilize electrophysiologic tests that are currently employed as clinical tests for endolymphatic hydrops. By using a combination of tests, evidence of hydrops will be sought in both the cochlea and the vestibular system.

1. Electrocochleography (ECoG). ECoG is an electrophysiologic test of cochlear function. Conditions such as Ménière's disease, which are characterized by endolymphatic hydrops, demonstrate an elevated summating potential to action potential (SP/AP) ratio on electrocochleography (ECoG). An increase in the SP relative to the AP is thought to be due to a deflection of the basilar membrane position toward the scala tympani. Accordingly, abnormal ECoG has been correlated with the finding of cochlear hydrops (in the basal turn) on gadolinium-enhanced MRI.
2. Vestibular evoked myogenic potentials (VEMPs). VEMPs arise from sound-induced activation of otolith organs and their associated vestibular neurons. The cervical VEMP (cVEMP) and ocular VEMP (oVEMP) are theorized to originate from the saccule and utricle, respectively. Thresholds, defined as the lowest stimulus intensity at which a response is seen, can be obtained at multiple test stimulus frequencies (250, 500, 750, 1000 Hz) and threshold response curves can be constructed. The lowest threshold for eliciting a response is typically seen at 500 Hz for both oVEMP and cVEMP. In hydropic conditions such as Ménière's disease, VEMP thresholds can be elevated or absent at all tested frequencies. Additionally, VEMP tuning curves can be shifted such that the lowest threshold is observed at a different tested frequency (e.g. 750 or 1000 Hz). A shift in resonance frequency of the otolithic organs due to pressure changes in the endolymphatic space is hypothesized to cause these changes.

Successful completion of the aims of this study will afford better understanding of the potential effects of infrasound on inner ear function. The findings of this work will fuel additional investigation of risks of infrasound exposure and may spur efforts to reduce individual and environmental exposure. A newly described mechanism would provide researchers, regulators and advocacy groups with a previously absent and crucial understanding of the effects of infrasound on inner ear function when crafting policy, designing new technologies, and ensuring the safety of exposed individuals

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 to 60 years
2. Absence of otologic symptoms based on screening questionnaire
3. Normal otoscopic examination
4. Audiometric thresholds less than 25 dB at 250, 500, 750, 1000 Hz.

Exclusion Criteria:

1. Age less than 18 or greater than 60 years. Age greater than 60 is considered an exclusion criterion as prior studies have demonstrated elevated VEMP thresholds attributed to age
2. Presence of any positive symptom on the questionnaire
3. Thresholds greater than 25 dB at the tested frequencies
4. Abnormal otoscopic examination (e.g., ear canal occlusion, tympanic membrane perforation, tympanic membrane retraction)
5. History of prior ear surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will be conducted in normal hearing adults. Each prospective participant will undergo a screening evaluation to determine eligibility, including: 1) completion of a basic otologic symptom questionnaire; 2) otoscopic examination; 3) binaural air conduction audiometry (250 to 1000 Hz).
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Measure the effects of infrasound exposure on the SP/AP ratio of electrocochleography | Test measurements at time -10, 10, and 20 minutes
  A baseline ECoG recording will be obtained and the waveform's SP/AP ratio will be calculated and recorded (time "-10"). A 10-minute infrasound stimulus will ensue. Immediately following cessation of the stimulus (time 10), a repeat ECoG test run will be performed. A 10-minute recovery period will take place followed by a final ECoG test run (time 20). S/P ratios will be recorded for each test run and percent change will be calculated.
Measure the effects of infrasound exposure on the threshold tuning curve of cVEMP | Test measurements at time -10, 10, and 20 minutes
  A baseline cVEMP tuning curve will be obtained and recorded (time "-10"). A 10-minute infrasound stimulus will ensue. Immediately following cessation of the stimulus (time 10), thresholds will be repeated. A 10-minute recovery period will take place followed by a final threshold measurement (time 20). Thresholds will be recorded for each test run and average change in threshold in dB will be calculated.
Measure the effects of infrasound exposure on the threshold tuning curve of oVEMP | Test measurements at time -10, 10, and 20 minutes
  A baseline oVEMP tuning curve will be obtained and recorded (time "-10"). A 10-minute infrasound stimulus will ensue. Immediately following cessation of the stimulus (time 10), thresholds will be repeated. A 10-minute recovery period will take place followed by a final threshold measurement (time 20). Thresholds will be recorded for each test run and average change in threshold in dB will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith E Adams, MD, Principal Investigator — Assistant Professor
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salt AN, Hullar TE. Responses of the ear to low frequency sounds, infrasound and wind turbines. Hear Res. 2010 Sep 1;268(1-2):12-21. doi: 10.1016/j.heares.2010.06.007. Epub 2010 Jun 16. PMID 20561575
- [Background] Berglund B, Hassmen P, Job RF. Sources and effects of low-frequency noise. J Acoust Soc Am. 1996 May;99(5):2985-3002. doi: 10.1121/1.414863. PMID 8642114
- [Background] Sugimoto T, Koyama K, Kurihara Y, Watanabe K. Measurement of infrasound generated by wind turbine generator. In: Proc. SICE Conf. 2008, pp. 5e8.
- [Background] Orrell A, Foster N. 2015 Distributed Wind Market Report. U.S. Department of Energy; 2016.
- [Background] Schmidt JH, Klokker M. Health effects related to wind turbine noise exposure: a systematic review. PLoS One. 2014 Dec 4;9(12):e114183. doi: 10.1371/journal.pone.0114183. eCollection 2014. PMID 25474326
- [Background] Kageyama T, Yano T, Kuwano S, Sueoka S, Tachibana H. Exposure-response relationship of wind turbine noise with self-reported symptoms of sleep and health problems: A nationwide socioacoustic survey in Japan. Noise Health. 2016 Mar-Apr;18(81):53-61. doi: 10.4103/1463-1741.178478. PMID 26960782
- [Background] May M, McMurtry RY. Wind Turbines and Adverse Health Effects: A Second Opinion. J Occup Environ Med. 2015 Oct;57(10):e130-2. doi: 10.1097/JOM.0000000000000447. No abstract available. PMID 26461874
- [Background] McCunney RJ, Mundt KA, Colby WD, Dobie R, Kaliski K, Blais M. Wind turbines and health: a critical review of the scientific literature. J Occup Environ Med. 2014 Nov;56(11):e108-30. doi: 10.1097/JOM.0000000000000313. PMID 25376420
- [Background] Flock A, Flock B. Hydrops in the cochlea can be induced by sound as well as by static pressure. Hear Res. 2000 Dec;150(1-2):175-88. doi: 10.1016/s0378-5955(00)00198-2. PMID 11077202
- [Background] Salt AN. Acute endolymphatic hydrops generated by exposure of the ear to nontraumatic low-frequency tones. J Assoc Res Otolaryngol. 2004 Jun;5(2):203-14. doi: 10.1007/s10162-003-4032-z. PMID 15357421
- [Background] Salt AN, Lichtenhan JT, Gill RM, Hartsock JJ. Large endolymphatic potentials from low-frequency and infrasonic tones in the guinea pig. J Acoust Soc Am. 2013 Mar;133(3):1561-71. doi: 10.1121/1.4789005. PMID 23464026
- [Background] Hensel J, Scholz G, Hurttig U, Mrowinski D, Janssen T. Impact of infrasound on the human cochlea. Hear Res. 2007 Nov;233(1-2):67-76. doi: 10.1016/j.heares.2007.07.004. Epub 2007 Jul 29. PMID 17761395
- [Background] Dommes E, Bauknecht HC, Scholz G, Rothemund Y, Hensel J, Klingebiel R. Auditory cortex stimulation by low-frequency tones-an fMRI study. Brain Res. 2009 Dec 22;1304:129-37. doi: 10.1016/j.brainres.2009.09.089. Epub 2009 Sep 28. PMID 19796632
- [Background] Coats AC. The summating potential and Meniere's disease. I. Summating potential amplitude in Meniere and non-Meniere ears. Arch Otolaryngol. 1981 Apr;107(4):199-208. doi: 10.1001/archotol.1981.00790400001001. PMID 7213179
- [Background] Durrant JD, Dallos P. Modification of DIF summating potential components by stimulus biasing. J Acoust Soc Am. 1974 Aug;56(2):562-70. doi: 10.1121/1.1903291. No abstract available. PMID 4414701
- [Background] Seo YJ, Kim J, Choi JY, Lee WS. Visualization of endolymphatic hydrops and correlation with audio-vestibular functional testing in patients with definite Meniere's disease. Auris Nasus Larynx. 2013 Apr;40(2):167-72. doi: 10.1016/j.anl.2012.07.009. Epub 2012 Aug 4. PMID 22867525
- [Background] Iwasaki S, Smulders YE, Burgess AM, McGarvie LA, Macdougall HG, Halmagyi GM, Curthoys IS. Ocular vestibular evoked myogenic potentials in response to bone-conducted vibration of the midline forehead at Fz. A new indicator of unilateral otolithic loss. Audiol Neurootol. 2008;13(6):396-404. doi: 10.1159/000148203. Epub 2008 Jul 29. PMID 18663292
- [Background] Rauch SD, Zhou G, Kujawa SG, Guinan JJ, Herrmann BS. Vestibular evoked myogenic potentials show altered tuning in patients with Meniere's disease. Otol Neurotol. 2004 May;25(3):333-8. doi: 10.1097/00129492-200405000-00022. PMID 15129114
- [Background] Winters SM, Berg IT, Grolman W, Klis SF. Ocular vestibular evoked myogenic potentials: frequency tuning to air-conducted acoustic stimuli in healthy subjects and Meniere's disease. Audiol Neurootol. 2012;17(1):12-9. doi: 10.1159/000324858. Epub 2011 Apr 29. PMID 21540585
- [Background] Koerner TK, Zhang Y, Nelson PB, Wang B, Zou H. Neural indices of phonemic discrimination and sentence-level speech intelligibility in quiet and noise: A mismatch negativity study. Hear Res. 2016 Sep;339:40-9. doi: 10.1016/j.heares.2016.06.001. Epub 2016 Jun 4. PMID 27267705
- [Background] Leventhall G. What is infrasound? Prog Biophys Mol Biol. 2007 Jan-Apr;93(1-3):130-7. doi: 10.1016/j.pbiomolbio.2006.07.006. Epub 2006 Aug 4. PMID 16934315
- [Background] Duck FA. Medical and non-medical protection standards for ultrasound and infrasound. Prog Biophys Mol Biol. 2007 Jan-Apr;93(1-3):176-91. doi: 10.1016/j.pbiomolbio.2006.07.008. Epub 2006 Aug 4. PMID 16965806
- [Background] Bonucci AS, Hyppolito MA. Comparison of the use of tympanic and extratympanic electrodes for electrocochleography. Laryngoscope. 2009 Mar;119(3):563-6. doi: 10.1002/lary.20105. PMID 19235755
- [Background] Densert B, Arlinger S, Sass K, Hergils L. Reproducibility of the electric response components in clinical electrocochleography. Audiology. 1994 Sep-Oct;33(5):254-63. doi: 10.3109/00206099409071885. PMID 7818379
- [Background] Blakley BW, Wong V. Normal Values for Cervical Vestibular-Evoked Myogenic Potentials. Otol Neurotol. 2015 Jul;36(6):1069-73. doi: 10.1097/MAO.0000000000000752. PMID 25839981
- [Background] Piker EG, Jacobson GP, McCaslin DL, Hood LJ. Normal characteristics of the ocular vestibular evoked myogenic potential. J Am Acad Audiol. 2011 Apr;22(4):222-30. doi: 10.3766/jaaa.22.4.5. PMID 21586257
- [Background] Adams ME, Heidenreich KD, Kileny PR. Audiovestibular testing in patients with Meniere's disease. Otolaryngol Clin North Am. 2010 Oct;43(5):995-1009. doi: 10.1016/j.otc.2010.05.008. PMID 20713239
- [Background] Janky KL, Shepard N. Vestibular evoked myogenic potential (VEMP) testing: normative threshold response curves and effects of age. J Am Acad Audiol. 2009 Sep;20(8):514-22. doi: 10.3766/jaaa.20.8.6. PMID 19764171